CLINICAL TRIAL: NCT06423872
Title: A Phase 1, Randomized, Parallel Assignment, Double Blind, Placebo Controlled, Single and Multiple Ascending Dose, Safety, Tolerability, and Pharmacokinetic Study of ZT002 in Healthy Participants
Brief Title: A SAD Study of ZT002 Injection in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing QL Biopharmaceutical Co.,Ltd (Industry)
Collaborators: Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BJQLZT002002
Record Dates: First submitted 2024-05-16; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ZT002 (Experimental): Participants will be randomized to receive ZT002 injection or Placebo in 1 of 6 dose cohorts.
  Interventions: Drug: ZT002
- Placebo (Placebo Comparator): Participants will be randomized to receive ZT002 injection or Placebo in 1 of 6 dose cohorts.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: ZT002 — Participants will receive a single subcutaneous (SC) ZT002 injection.
  Arms: ZT002
Other: Placebo — Participants will receive same volume as of the study drug.
  Arms: Placebo

SUMMARY:
This study will comprise a randomized, parallel assignment, double blind, placebo controlled, single and multiple ascending dose, safety, tolerability and pharmacokinetic study of ZT002 in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the purpose, nature, methods, and potential adverse reactions of the experiment, voluntarily participate as a participant, comply with the requirements of this study, and sign an informed consent form.
2. Healthy adults, age 18~45 years, both inclusive, at time of informed consent.
3. Body Mass Index (BMI) between 19～27.0 kg/m2 both included. Male weight>55.0kg, famale weight>50.0kg.
4. In good health, determined by no clinically significant findings from medical history, physical examination, vital signs measurements, anterior and lateral chest X-ray,12-lead ECG, and clinical laboratory evaluations(blood routine, blood biochemistry, coagulation function, and urine routine)at screening and before administration of study drug, as assessed by the Investigator.
5. Female participants are required to abstain or use two effective contraceptive methods simultaneously from 1 month before screening to 6 months after the last dose. Male participants are required to abstain or use two effective contraceptive methods simultaneously from the first dose to 6 months after the last dose: male participants are required to undergo surgical sterilization (such as vas deferens ligation) or use condoms correctly, or their spouse is required to use hormonal contraceptives approved by the National Medical Products Administration (such as contraceptive pills, patches, implantable or injectable preparations) or intrauterine devices (IUDs) or undergo surgical sterilization; Female subjects may undergo surgical sterilization (such as tubal ligation) or intrauterine devices (IUDs), or their spouses may use condoms correctly or undergo surgical sterilization. After the trial, female subjects may also use hormone contraceptives approved by the National Medical Products Administration (such as contraceptive pills, patches, implantable or injectable preparations).

Exclusion Criteria:

1. History of drug allergy or allergic related diseases (allergic rhinitis, asthma, urticaria, eczema, etc.)，allergic to experimental drugs and excipients or GLP-1 class drugs.
2. Significant history or clinical manifestation of any neurological, cardiovascular, hematological, hepatic, renal, gastrointestinal, respiratory, metabolic, endocrine, immune or skeletal, as determined by the Investigator.
3. Family or personal history of medullary thyroid carcinoma (MTC).
4. Medical history of multiple endocrine neoplasia type 2(MEN2).
5. History of acute or chronic pancreatitis.
6. History of hypoglycemia.
7. Calcitonin equal or above 50 ng/L at screening.
8. The content of amylase or lipase during the screening period is higher than the upper limit of normal values and has clinical significance.
9. Screening period HbAlc (glycated hemoglobin) ≥ 6.5%.
10. According to the Fridericias formula，QTcF ≥ 450 ms for subjects in 12-lead ECG examination during screening or baseline period.
11. History of drug abuse within the previous year of screening or positive results from drug abuse screening (urine screening).
12. Have smoked ≥5 cigarettes per day in the past 3 month prior to Screening or unable to refrain from smoking during the study.
13. Screening for subjects who have consumed more than 14 units of alcohol per week within the first 3 months (1 unit of alcohol=360 mL of beer or 45 mL of 40% alcohol or 150 mL of wine), or who have taken alcoholic products within 48 hours before administration, or who cannot abstain from alcohol during the trial period.
14. Positive test for hepatitis B surface antigen (HBsAg)，hepatitis C antibody (HCV-Ab), human immunodeficiency virus (HIV-Ab) antibody, treponema pallidum(TP-Ab) antibody at screening.
15. Screening for subjects who have participated in other clinical trials and received drug therapy or medical device intervention within the first 3 months.
16. Blood donation or blood loss - more than 400 mL during the 3 months prior to screening, or received blood transfusion; or blood donation or blood loss - more than 200 mL during the 1 months prior to screening.
17. History of infectious diseases within 4 weeks before screening (judged by the investigator to affect the ability of the subject to participate in the test)
18. Cannot tolerate venous puncture blood collection or have a history of fainting or fainting
19. Received vaccination within 28 days prior to administration or plan to receive vaccination during the study period.
20. Use of prescription or non-prescription or chinese herbal medicine or discontinue medication before 1 month to screening or within 5 half-lives of the medicinal product, (whichever is longest).
21. Participant is unable to refrain from strenuous exercise during the study
22. Breastfeeding or pregnant women, or positive tests of pregnancy in screening or baseline
23. Other unsuitable conditions to participate in the clinical study judged by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-12-08 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of a single escalation dose of ZT002 through the incidence and severity of treatment emergent adverse events in SAD Cohorts. Number of participants with treatment-emergent adverse events | Up to 50 days
  Coded by the most updated version of the Medical Dictionary for Regulatory Activities (MedDRA).
Safety and tolerability of a single escalation dose of ZT002 through the incidence severity of serious adverse events in SAD Cohorts. Number of participants with serious adverse events. | Up to 50 days
  Coded by the most updated version of the Medical Dictionary for Regulatory Activities (MedDRA).

SECONDARY OUTCOMES:
The Pharmacokinetics (PK) profile of a single escalation dose of ZT002 in healthy participants in SAD Cohorts. | Up to 50 days
  Parameter: Maximum observed plasma concentration of ZT002 (Cmax)
The Pharmacokinetics (PK) profile of a single escalation dose of ZT002 in healthy participants in SAD Cohorts. | Up to 50 days
  Parameter: Area under the drug-time curve from 0 h after dosing to the last quantifiable concentration time point (AUC0-last)
The Pharmacokinetics (PK) profile of a single escalation dose of ZT002 in healthy participants in SAD cohorts. | Up to 50 days
  Parameter: Area under the drug-time curve to infinity (AUC0-inf)

CONTACTS AND LOCATIONS:
Overall Officials: Aixin Shi, Master, Principal Investigator — No.1 Dahua Road, Dongdan, Dongcheng District, Beijing
Locations (1):
- Beijing Hospital, Beijing, Beijing Municipality, China